CLINICAL TRIAL: NCT03968978
Title: A Multicenter, Randomized, Open-label, Parallel Group, Functionality, and Performance Study of an Accessorized Pre-filled Syringe and Autoinjector With Home-administered Subcutaneous Tezepelumab in Adolescent and Adult Subjects With Severe Asthma (PATH-HOME)
Brief Title: Tezepelumab Home Use Study
Acronym: PATH-HOME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5180C00011
Record Dates: First submitted 2019-04-30; First posted 2019-05-30 (Actual); Results first posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Asthma
Keywords: Asthma, Severe Uncontrolled Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to either an accessorized pre-filled syringe or an autoinjector. Both will be administered 210 mg tezepelumab subcutaneously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tezepelumab (AI) (Experimental): Tezepelumab subcutaneous injection, administered by Autoinjector (AI) device.
  Interventions: Biological: Tezepelumab (AI)
- Tezepelumab (APFS) (Experimental): Tezepelumab subcutaneous injection, administered by Accessorized pre-filled syringe (APFS).
  Interventions: Biological: Tezepelumab (APFS)

INTERVENTIONS:
Biological: Tezepelumab (APFS) — Tezepelumab subcutaneous injection, administered by Accessorized pre-filled syringe (APFS).
  Arms: Tezepelumab (APFS)
Biological: Tezepelumab (AI) — Tezepelumab subcutaneous injection, administered by Autoinjector (AI) device.
  Arms: Tezepelumab (AI)

SUMMARY:
This is a multicenter, randomized, open-label, parallel-group study designed to assess healthcare provider and subject/caregiver reported functionality and performance of a single-use accessorized pre-filled syringe (APFS) or autoinjector (AI) with a fixed 210 mg dose of tezepelumab administered subcutaneously in the clinic and in an at-home setting.

DETAILED DESCRIPTION:
The study will consist of a screening/run-in period of up to 2 weeks and a treatment period of 24 weeks, followed by a post-treatment follow-up period of 12 weeks. During the treatment period, one dose of 210 mg tezepelumab will be administered via a single-use APFS or AI subcutaneously (SC) every 4 weeks (Q4W) starting at Visit 2 (Week 0) until Visit 7 (Week 20). Subjects will be administered tezepelumab at the site during Visits 2 (Week 0), 3 (Week 4), 4 (Week 8) and 7 (Week 20). At-home administration of tezepelumab will occur during Visit 5 (Week 12) and Visit 6 (Week 16). Each device will be assessed separately using descriptive presentations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 12 to 80 years.
* Documented physician-diagnosed asthma for at least 12 months.
* Evidence of asthma as documented by post BD (albuterol/salbutamol) reversibility of FEV1 ≥ 12% AND ≥200 mL (15-60 min after administration of 4 puffs of albuterol/salbutamol), documented either: in the previous 12 months prior to V1, OR demonstrated at V1, V1A, or at V2.
* Documented history of current treatment with medium- or high-dose ICS for at least 6 months and at least one additional asthma controller medication according to standard practice of care. ICS dose must be greater than or equal to 500 μg/day fluticasone propionate dry powder formulation or equivalent daily.
* Morning pre-BD FEV1 of >50% predicted normal at Visit 1, Visit 1A, or Visit 2.

Exclusion Criteria:

* Clinically important pulmonary or systemic diseases other than asthma.
* History of cancer except basal cell carcinoma, squamous cell carcinoma, or in situ carcinoma of the cervix within 12 months prior to Visit 1.
* Acute upper or lower respiratory infection requiring antibiotics or antiviral medications finalized <2 weeks before Visit 1 or during screening/run-in period.
* A helminth parasitic infection diagnosed within 6 months that is untreated or is unresponsive to the standard of care.
* Smoking history of ≥10 pack years, (includes vaping and e-cigarettes)
* History of chronic alcohol or drug abuse.
* Tuberculosis requiring treatment within 12 months prior to V1.
* History of HIV, Hepatitis B or Hepatitis C.
* Receipt of any marketed or investigational biologic agent within 4 months or 5 half-lives (whichever is longer) prior to visit 1 or receipt of any investigational non-biologic agent within 30 days or 5 half-lives.
* Bronchial thermoplasty in 24 months prior to V1.
* Anaphylaxis or documented immune complex disease (Type III hypersensitivity reactions) to any biologic therapy.
* Evidence of active liver disease (e.g. jaundice, AST, ALT or ALP >2 times upper limit of normal), ongoing liver disease or inexplicably elevated liver chemistry values.
* Pregnant, breastfeeding or lactating women.
* Non-leukocyte depleted whole blood transfusion in 120 days prior to visit 1.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sady A Alpizar, MD, Principal Investigator — Clinical Research Trials of Florida, Inc.
Locations (33):
- United States (15):
  - Research Site, Hoover, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Northridge, California
  - Research Site, Palm Desert, California
  - Research Site, Westminster, California
  - Research Site, Tampa, Florida
  - Research Site, Savannah, Georgia
  - Research Site, Omaha, Nebraska
  - Research Site, Northfield, New Jersey
  - Research Site, Cincinnati, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Dallas, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
- Canada (9):
  - Research Site, Calgary, Alberta
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Fukuoka
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Strzelce Opolskie
  - Research Site, Tarnów
  - Research Site, Wieluń
  - Research Site, Wroclaw

REFERENCES:
- [Derived] Alpizar S, Megally A, Chen C, Raj A, Downie J, Colice G. Functionality and Performance of an Accessorized Pre-Filled Syringe and an Autoinjector for At-Home Administration of Tezepelumab in Patients with Severe, Uncontrolled Asthma. J Asthma Allergy. 2021 Apr 19;14:381-392. doi: 10.2147/JAA.S305114. eCollection 2021. PMID 33907423
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00011&attachmentIdentifier=34dcbdad-0c68-4350-8ed5-7194d8bb9c97&fileName=D5180C00011-sap-ed-2_(03-Sep-2020)-redacted.pdf&versionIdentifier=
- See also: Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00011&attachmentIdentifier=35e421e0-5181-469c-a1b9-577eb9e0d37b&fileName=D5180C00011-csp-v2_-_CI_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 216 subjects randomized in the study.
Pre-assignment Details: 216 subjects randomized to tezepelumab 210 mg Q4W via APFS and tezepelumab 210 mg Q4W via AI. All randomized subjects were treated. 111 (51.4%) were randomized to tezepelumab 210 mg Q4W via APFS and 105 (48.6%) were randomized to tezepelumab 210 mg Q4W via AI.
Groups:
- Teze 210 mg Q4W Via APFS: Accessorized pre-filled syringe every 4 weeks administered subcutaneously
- Teze 210 mg Q4W Via AI: Autoinjector every 4 weeks administered subcutaneously
Period: Overall Study
Arm/Group | Teze 210 mg Q4W Via APFS | Teze 210 mg Q4W Via AI
Started | 111 | 105
Completed | 110 | 105
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teze 210 mg Q4W Via APFS | Teze 210 mg Q4W Via AI | Total
Number analyzed (Participants) | 111 | 105 | 216
Age, Continuous [Mean (Standard Deviation); unit: Years] — Measure analysis population description for: Full Analysis Set
  Years | 48.5 (18.1) | 45.8 (18.3) | 47.2 (18.2)
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (>=12 to <18 years) | 13 | 11 | 24
  Adults (>=18 years) | 98 | 94 | 192
  Adults (>=18 to <65 years) | 79 | 73 | 152
  Adults (>=65 years) | 19 | 21 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 52 | 108
  Male | 55 | 53 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 87 | 82 | 169
  Black or African American | 8 | 8 | 16
  Asian | 16 | 15 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 99 | 92 | 191

OUTCOME MEASURES:

1. Primary Outcome: Proportions of HCPs and Subjects/Caregivers Who Successfully Administered Tezepelumab in Clinic or at Home by Device Type
Description: Successful administration is defined as an injection completed, based on a used/returned (HCP or subject/caregiver) answer of YES to all 5 questions in the administration questionnaire, and satisfactory in vitro evaluation of returned/evaluated devices.
Time Frame: Week 0, Week 4, Week 8, Week 12, Week 16, Week 20
Population: Full analysis set - Include all subjects randomised to study treatment who received or attempted to receive at least one dose of investigational product, irrespective of their protocol adherence and continued participation.
Measure: Count of Participants; unit: Participants
Arm/Group | Teze 210 mg Q4W Via APFS | Teze 210 mg Q4W Via AI
Number analyzed (Participants) | 111 | 105
Participants
  Week 0 (in clinic) | 109 | 105
  Week 4 (in clinic) | 111 | 102
  Week 8 (in clinic): number analyzed (Participants) | 110 | 105
  Week 8 (in clinic) | 110 | 103
  Week 12 (at home): number analyzed (Participants) | 110 | 105
  Week 12 (at home) | 110 | 104
  Week 16 (at home): number analyzed (Participants) | 109 | 105
  Week 16 (at home) | 104 | 102
  Week 20 (in clinic): number analyzed (Participants) | 109 | 105
  Week 20 (in clinic) | 105 | 102
Statistical Analysis 1: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI at Week 0 (in clinic); Proportion = 98.2, 95% CI 2-sided [93.67 to 99.5]
Statistical Analysis 2: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI at Week 4 (in clinic); Proportion = 100, 95% CI 2-sided [96.65 to 100]
Statistical Analysis 3: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI for Week 8 (in clinic); Proportion = 100.0, 95% CI 2-sided [96.63 to 100.00]
Statistical Analysis 4: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI for Week 12 (at home); Proportion = 100.0, 95% CI 2-sided [96.63 to 100.00]
Statistical Analysis 5: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI for Week 16 (at home); Proportion = 95.4, 95% CI 2-sided [89.71 to 98.02]
Statistical Analysis 6: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI for Week 20 (in clinic); Proportion = 96.3, 95% CI 2-sided [90.94 to 98.56]
Statistical Analysis 7: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for Week 0 (in clinic); Proportion = 100.0, 95% CI 2-sided [96.47 to 100.00]
Statistical Analysis 8: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for Week 4 (in clinic); Proportion = 97.1, 95% CI 2-sided [91.93 to 99.02]
Statistical Analysis 9: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for Week 8 (in clinic); Proportion = 98.1, 95% CI 2-sided [93.32 to 99.48]
Statistical Analysis 10: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for week 12 (at home); Proportion = 99.0, 95% CI 2-sided [94.80 to 99.83]
Statistical Analysis 11: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for Week 16 (at home); Proportion = 97.1, 95% CI 2-sided [91.93 to 99.02]
Statistical Analysis 12: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for Week 20 (in clinic); Proportion = 97.1, 95% CI 2-sided [91.93 to 99.02]

2. Secondary Outcome: Proportions of Used/Returned Devices That Pass Functional Tests and Visual Inspection and Showed no Evidence of Malfunction
Description: Devices that passed functional tests and visual inspection and showed no evidence of malfunction will be evaluated as functional.
  Percentages have been calculated by using the number of used and returned devices at specified visit as denominator.
  Note: A few participants had missing devices. One participant had two AI devices at Week 4.
Time Frame: Week 0, Week 4, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 1
Measure: Count of Units; unit: Devices
Units Other Than Participants: Devices
Arm/Group | Teze 210 mg Q4W Via APFS | Teze 210 mg Q4W Via AI
Number analyzed (Participants) | 111 | 105
Number analyzed (Devices) | 655 | 624
Devices
  Week 0 (in clinic): number analyzed (Devices) | 111 | 105
  Week 0 (in clinic) | 109 | 105
  Week 4 (in clinic): number analyzed (Devices) | 111 | 106
  Week 4 (in clinic) | 111 | 103
  Week 8 (in clinic): number analyzed (Devices) | 110 | 105
  Week 8 (in clinic) | 110 | 103
  Week 12 (at home): number analyzed (Devices) | 110 | 104
  Week 12 (at home) | 110 | 104
  Week 16 (at home): number analyzed (Devices) | 107 | 102
  Week 16 (at home) | 104 | 102
  Week 20 (in clinic): number analyzed (Devices) | 106 | 102
  Week 20 (in clinic) | 105 | 102
Statistical Analysis 1: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI at Week 0 (in clinic); Proportion = 98.2, 95% CI 2-sided [93.67 to 99.50]
Statistical Analysis 2: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI at Week 4 (in clinic); Proportion = 100.0, 95% CI 2-sided [96.65 to 100.00]
Statistical Analysis 3: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI for Week 8 (in clinic); Proportion = 100.0, 95% CI 2-sided [96.63 to 100.00]
Statistical Analysis 4: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI for Week 12 (at home); Proportion = 100.0, 95% CI 2-sided [96.63 to 100.00]
Statistical Analysis 5: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI for Week 16 (at home); Proportion = 97.2, 95% CI 2-sided [92.80 to 99.04]
Statistical Analysis 6: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI for Week 20 (in clinic); Proportion = 99.1, 95% CI 2-sided [94.85 to 99.83]
Statistical Analysis 7: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for Week 0 (in clinic); Proportion = 100.0, 95% CI 2-sided [96.46 to 100.00]
Statistical Analysis 8: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for Week 4 (in clinic); Proportion = 97.2, 95% CI 2-sided [93.38 to 99.48]
Statistical Analysis 9: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Other CI; CI for Week 8 (in clinic); Proportion = 98.1, 95% CI 2-sided [93.32 to 99.48]
Statistical Analysis 10: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for week 12 (at home); Proportion = 100.0, 95% CI 2-sided [96.44 to 100.00]
Statistical Analysis 11: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for Week 16 (at home); Proportion = 100.0, 95% CI 2-sided [96.37 to 100.00]
Statistical Analysis 12: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for Week 20 (in clinic); Proportion = 100.0, 95% CI 2-sided [96.37 to 100.00]

3. Secondary Outcome: Proportions of Devices That Have Been Reported as Malfunctioning (Product Complaints)
Description: Performance is measured by the proportion of APFS or AI devices that have been reported as malfunctioning (i.e. via Product Complaints).
  Percentages have been calculated by using the number of used and returned devices at specified visit as denominator.
  Note: A few participants had missing devices. One participant had two AI devices at Week 4.
Time Frame: Week 0, Week 4, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 1
Measure: Count of Units; unit: Devices
Units Other Than Participants: Devices
Arm/Group | Teze 210 mg Q4W Via APFS | Teze 210 mg Q4W Via AI
Number analyzed (Participants) | 111 | 105
Number analyzed (Devices) | 655 | 624
Devices
  Week 0 (in clinic): number analyzed (Devices) | 111 | 105
  Week 0 (in clinic) | 2 | 0
  Week 4 (in clinic): number analyzed (Devices) | 111 | 106
  Week 4 (in clinic) | 0 | 3
  Week 8 (in clinic): number analyzed (Participants) | 110 | 105
  Week 8 (in clinic): number analyzed (Devices) | 110 | 105
  Week 8 (in clinic) | 0 | 2
  Week 12 (at home): number analyzed (Participants) | 110 | 104
  Week 12 (at home): number analyzed (Devices) | 110 | 104
  Week 12 (at home) | 0 | 0
  Week 16 (at home): number analyzed (Participants) | 107 | 102
  Week 16 (at home): number analyzed (Devices) | 107 | 102
  Week 16 (at home) | 3 | 0
  Week 20 (in clinic): number analyzed (Participants) | 106 | 102
  Week 20 (in clinic): number analyzed (Devices) | 106 | 102
  Week 20 (in clinic) | 1 | 0
Statistical Analysis 1: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI at Week 0 (in clinic); Proportion = 1.8, 95% CI 2-sided [0.50 to 6.33]
Statistical Analysis 2: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI at Week 4 (in clinic); Proportion = 0, 95% CI 2-sided [0 to 3.35]
Statistical Analysis 3: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI for Week 8 (in clinic); Proportion = 0, 95% CI 2-sided [0 to 3.37]
Statistical Analysis 4: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI for Week 12 (at home); Proportion = 0, 95% CI 2-sided [0 to 3.37]
Statistical Analysis 5: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI for Week 16 (at home); Proportion = 2.8, 95% CI 2-sided [0.96 to 7.92]
Statistical Analysis 6: Comparison: Teze 210 mg Q4W Via APFS; Test type: Other; Score CI; CI for Week 20 (in clinic); Proportion = 0.9, 95% CI 2-sided [0.17 to 5.15]
Statistical Analysis 7: Comparison: Teze 210 mg Q4W Via AI; Test type: Superiority; Score CI; CI for Week 0 (in clinic); Proportion = 0, 95% CI 2-sided [0 to 3.53]
Statistical Analysis 8: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for Week 4 (in clinic); Proportion = 2.8, 95% CI 2-sided [0.97 to 7.99]
Statistical Analysis 9: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Other CI; CI for Week 8 (in clinic); Proportion = 1.9, 95% CI 2-sided [0.52 to 6.68]
Statistical Analysis 10: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for week 12 (at home); Proportion = 0, 95% CI 2-sided [0 to 3.56]
Statistical Analysis 11: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for Week 16 (at home); Proportion = 0, 95% CI 2-sided [0 to 3.63]
Statistical Analysis 12: Comparison: Teze 210 mg Q4W Via AI; Test type: Other; Score CI; CI for Week 20 (in clinic); Proportion = 0, 95% CI 2-sided [0 to 3.63]

4. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-6 (ACQ-6) Score
Description: The ACQ-6 captures asthma symptoms and short-acting β2-agonist use via subject-report. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The ACQ-6 score is the mean of the responses.
Time Frame: Baseline (Week 0), Week 4, Week 8, Week 12, Week 16, Week 20 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Teze 210 mg Q4W Via APFS | Teze 210 mg Q4W Via AI
Number analyzed (Participants) | 111 | 105
Score
  ACQ-6 score at Baseline (Week 0) | 2.227 (0.732) | 2.081 (0.625)
  ACQ-6 score at Week 4 | 1.629 (0.791) | 1.492 (0.715)
  Change from Baseline of ACQ-6 score at Week 4 | -0.598 (0.702) | -0.589 (0.694)
  ACQ-6 score at Week 8 | 1.401 (0.859) | 1.316 (0.744)
  Change from Baseline of ACQ-6 score at Week 8 | -0.826 (0.833) | -0.765 (0.793)
  ACQ-6 score at Week 12: number analyzed (Participants) | 110 | 105
  ACQ-6 score at Week 12 | 1.197 (0.751) | 1.143 (0.745)
  Change from Baseline of ACQ-6 score at Week 12: number analyzed (Participants) | 110 | 105
  Change from Baseline of ACQ-6 score at Week 12 | -1.011 (0.805) | -0.938 (0.805)
  ACQ-6 score at Week 16: number analyzed (Participants) | 109 | 105
  ACQ-6 score at Week 16 | 1.226 (0.845) | 1.171 (0.782)
  Change from Baseline of ACQ-6 score at Week 16: number analyzed (Participants) | 109 | 105
  Change from Baseline of ACQ-6 score at Week 16 | -0.986 (0.893) | -0.910 (0.867)
  ACQ-6 score at Week 20: number analyzed (Participants) | 108 | 105
  ACQ-6 score at Week 20 | 1.230 (0.832) | 1.238 (0.795)
  Change from Baseline of ACQ-6 score at Week 20: number analyzed (Participants) | 108 | 105
  Change from Baseline of ACQ-6 score at Week 20 | -0.978 (0.866) | -0.843 (0.910)
  ACQ-6 score at Week 24: number analyzed (Participants) | 109 | 105
  ACQ-6 score at Week 24 | 1.072 (0.755) | 1.140 (0.765)
  Change from Baseline of ACQ-6 score at Week 24: number analyzed (Participants) | 109 | 105
  Change from Baseline of ACQ-6 score at Week 24 | -1.141 (0.845) | -0.941 (0.775)

5. Secondary Outcome: Serum Trough Concentrations
Description: PK serum samples were collected pre-dose on dosing visits
Time Frame: Baseline (Week 0), Week 4, Week 20 and Week 24 (EOT)
Population: PK analysis set - Includes all subjects in the full analysis set who received tezepelumab treatment and had at least one sample with one detectable serum concentration from a sample collected post-treatment that is assumed not to be affected by factors such as protocol deviations (e.g. disallowed medication or incorrect study medication received).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Teze 210 mg Q4W Via APFS | Teze 210 mg Q4W Via AI
Number analyzed (Participants) | 111 | 105
µg/mL
  Baseline (Week 0) | NA (NA) — <LLOQ (Lower Limit of Quantification) | NA (NA) — <LLOQ (Lower Limit of Quantification)
  Week 4: number analyzed (Participants) | 109 | 105
  Week 4 | 10.9764 (48.3948) | 10.5690 (57.0076)
  Week 20: number analyzed (Participants) | 108 | 105
  Week 20 | 18.9653 (69.0785) | 20.3206 (56.5858)
  Week 24 (EOT): number analyzed (Participants) | 109 | 105
  Week 24 (EOT) | 19.6274 (58.2660) | 19.9264 (54.3198)

6. Secondary Outcome: Anti-drug Antibodies (ADA)
Description: Anti-drug antibodies (ADA) responses at baseline and/or post baseline. Treatment-induced ADA positive is defined as ADA negative at baseline and post-baseline ADA positive. Treatment-boosted ADA positive is defined as baseline positive ADA titre that was boosted to a 4-fold or higher-level following IP administration. Treatment-emergent ADA (TE-ADA) positive is defined as either treatment-induced ADA positive or treatment-boosted ADA positive. ADA incidence is the proportion of TE-ADA positive subjects in a population. Persistently positive is defined as ADA positive at >=2 post-baseline assessments (with >=16 weeks between first and last positive) or ADA positive at last post-baseline assessment. Transiently positive is defined as having at least one post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive
Time Frame: Pre-treatment on dosing days until end of follow-up (Week 36) per protocol
Population: Safety analysis set - Includes all subjects who received at least one dose of tezepelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Teze 210 mg Q4W Via APFS | Teze 210 mg Q4W Via AI
Number analyzed (Participants) | 111 | 105
Participants
  ADA positive at baseline and/or post-baseline (ADA prevalence) | 2 | 11
  TE-ADA positive (ADA incidence) | 2 | 8
  Treatment-induced ADA positive | 2 | 8
  Treatment-boosted ADA positive | 0 | 0
  ADA persistently positive | 1 | 7
  ADA transiently positive | 1 | 3
  Only baseline ADA positive | 0 | 1
  Both baseline and at least one post-baseline ADA positive | 0 | 2

ADVERSE EVENTS:
Time Frame: From first dose till end of study (Week 36)
Arm/Group | Teze 210 mg Q4W Via APFS | Teze 210 mg Q4W Via AI
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/105
Serious Adverse Events (participants affected / at risk) | 5/111 | 4/105
Other Adverse Events (participants affected / at risk) | 29/111 | 29/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teze 210 mg Q4W Via APFS (N=111) | Teze 210 mg Q4W Via AI (N=105)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Genitourinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Psychogenic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teze 210 mg Q4W Via APFS (N=111) | Teze 210 mg Q4W Via AI (N=105)
Nasopharyngitis (Infections and infestations) | 12 (13) | 15 (15)
Pharyngitis (Infections and infestations) | 4 (4) | 4 (6)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 8 (9)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT03968978/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT03968978/SAP_001.pdf